CLINICAL TRIAL: NCT06516042
Title: Effectiveness, Feasibility, and Acceptability of Targeted Antimalarial Interventions for Seasonal Migrant Populations in Metema District, Amhara Region, Ethiopia
Brief Title: Targeted Antimalarial Drug Administration for Seasonal Migrant Populations in Amhara Region, Ethiopia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Federal Minstry of Health of Ethiopia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RES-00764
Record Dates: First submitted 2024-07-11; First posted 2024-07-23 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Plasmodium Falciparum; Malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — piperaquine; artenimol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention with 2 TDA rounds (Active Comparator): TDA with DP will be administered two times with a 4 - 6 week interval between rounds to all workers in the selected farm sites
  Interventions: Drug: Dihydroartemisinin-piperaquine
- Intervention with 3 TDA rounds (Active Comparator): TDA with DP will be administered three times with a 4 - 6 week interval between rounds to all workers in the selected farm sites
  Interventions: Drug: Dihydroartemisinin-piperaquine
- Control (no TDA) (No Intervention): TDA with DP will not be administered to any workers in the selected farm sites

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — Participants that provide consent to participate in the TDA and are deemed eligible for treatment will receive a course of dihydroartemisinin-piperaquine (DP) if male, and artemether-lumefantrine (AL) if female. They will take the first dose of the treatment under direct observed therapy, and will receive the rest of the tablets to take on their own for days two and three.
  Other Names: Piperaquine/dihydroartemisinin
  Arms: Intervention with 2 TDA rounds; Intervention with 3 TDA rounds

SUMMARY:
The purpose of the study is to assess the effectiveness, feasibility, and acceptability of targeted drug administration for seasonal migrant populations in Metema District, Amhara Region, Ethiopia

DETAILED DESCRIPTION:
A cluster randomized controlled trial will be used to evaluate the effectiveness, feasibility, and acceptability of targeted antimalarial drug administration (TDA) for seasonal migrant farmworkers in the Delello farm sites in Metema district, Amhara Region. Individual farm sites will be randomized 1:1:1 to either of two intervention options or control, where all farmworkers at intervention sites will receive either two or three rounds of dihydro artemisinin piperaquine over the primary farming season.

All study farm-sites will receive enhanced case management conducted by mobile health teams throughout the study period.

Cross-sectional surveys will be conducted in all arms at baseline and 4 to 6 weeks following the third round of TDA to assess the effectiveness of the intervention for reducing parasite prevalence.

ELIGIBILITY:
Inclusion Criteria:

* At the time of the study, be a seasonal farm worker at one of the selected farm sites in Metema district
* Available and willingness to participate in the study and provide consent (or parental/guardian consent and asset in the case of minors)

Exclusion Criteria:

* Severe illness (will be referred for care)
* Inability to provide informed consent
* Age 14-17 years old and not having a parent/guardian at the farm who can provide consent
* Age <14 years old

Additional exclusion criteria for the intervention group:

* Having received an antimalarial drug within the last 2 weeks
* Having any of the contraindications to receiving DP:

  * History of cardiac rhythm disturbances, bradycardia, or heart failure
  * Concomitant treatment with drugs that prolong the QT interval (fluconazole, fluoroquinolones, hydroxyzine, macrolides, ondansetron, etc.) or drugs containing any of the following: flecainide, metoprolol, imipramine, amitriptyline, clomipramine
  * Known allergic reactions to DP or other artemisinin derivatives
  * Pregnancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10350 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Plasmodium falciparum (Pf) parasite prevalence | Up to 6 months
  Prevalence of Pf as determined by PCR at the end of the study
Feasibility of TDA | Up to 6 months
  Feasibility of TDA measured through intervention coverage (% of participants treated among the total farm population) and cost effectiveness
Acceptability of TDA amongst farmworkers, farm-site owners, and local health authorities | Up to 6 months
  Acceptability of TDA amongst farmworkers, farm-site owners, and local health authorities measured through drug adherence (% of participants completing the drugs as prescribed, as reported in the endline survey), survey response (self-reported values provided during endline survey), and qualitative interview data

SECONDARY OUTCOMES:
Pf parasite prevalence in a subset of migrant farmworkers | Up to 2 months
  Pf parasite prevalence measured in a subset of migrant farmworkers upon return to their home village in the western highlands
Safety and tolerability of TDA | Up to 6 months
  Safety and tolerability of TDA measured through the incidence of adverse events and survey responses
Feasibility of enhanced case management through mobile clinics based on cost per case detected | Up to 6 months
  A cost assessment of providing enhanced case management through mobile clinics
Feasibility and acceptability of enhanced case management through mobile clinics based on endline survey responses | Up to 6 months
  Feasibility and acceptability of providing enhanced case management among the study team based on endline survey responses
Feasibility and acceptability of enhanced case management through mobile clinics based on qualitative interview data | Up to 6 months
  Feasibility and acceptability of enhanced case management through mobile clinics based on information shared during qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bennett, PhD, Principal Investigator — PATH; Henry Ntuku, MD, PhD, Principal Investigator — PATH; Gudissa Assefa Bayissa, Principal Investigator — Ethiopia Federal Ministry of Health; Hiwot Teka, Principal Investigator — President's Malaria Initiative
Locations (1):
- Delello Farm Sites, Gonder, Metema District, Ethiopia

IPD SHARING:
Plan to Share IPD: No
For all data collected as part of the study, participants will be assigned a unique identification number. Individual identifiers (names, cell phone number) will be collected to support any follow up if needed. However, no personal identification information will be used in any reports arising out of this research.
  Dried blood spots (DBS) will be collected from participants and shared with the Armauer Hansen Research Institute for sample analysis and storage. Stored biospecimens will be deidentified with no possibility of linking with study participants. Only a unique sample identification code will identify the samples. Results might be linked to the associated epidemiological data collected during the surveys from the participants, which will not include any identifiable information.